CLINICAL TRIAL: NCT03101943
Title: Preventing Early Childhood Obesity, Part 1: Family Spirit Nurture, 3-9 Months
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7476
Record Dates: First submitted 2017-02-20; First posted 2017-04-05 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Obesity; Water; Lack of; Breast Feeding; Tooth Erosion; Dental Plaque; Infant Obesity; Feeding Behavior; Mother-Child Relations; Dietary Habits; Dental Caries
Keywords: Sugar; Sweetened; Beverages
MeSH Terms: conditions — Obesity; Breast Feeding; Tooth Erosion; Dental Plaque; Pediatric Obesity; Feeding Behavior; Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Spirit Nurture (FSN) (Experimental): The intervention group (n=68) will receive the Family Spirit Nurture (FSN) home-visiting module, consisting of six 45-minute lessons delivered biweekly by trained local American Indian Family Health Coaches (FHCs), from 3 to 6 months postpartum. The lessons focus on elimination or reduction of Sugar Sweetened Beverages (SSBs) among infants while teaching mothers complementary feeding and responsive parenting practices. Lessons are highly visual and interactive, and will incorporate cultural teachings related to infant feeding and nutrition that support aims. All families will receive water delivery of drinking water from 6 to 9 months postpartum.
  Interventions: Behavioral: Family Spirit Nurture (FSN); Other: Water Delivery
- Control Program (Other): The control group (n=68) will receive three home-based lessons with home safety information (injury prevention is a priority identified by Navajo leadership that does not interfere with study questions). Mothers randomized to the control group will receive 3 educational lessons on home safety and child safety proofing. These meaningful topics were selected so as not to dilute measurement on key FSN outcomes and to provide benefit to all study participants. Lessons will be delivered monthly (at 3, 4 and 5 months postpartum) in the same format as the FSN lessons, by trained FHCs in the home of the participant or in a private place of their choosing. All families will receive water delivery of drinking water from 6 to 9 months postpartum.
  Interventions: Other: Control Program; Other: Water Delivery

INTERVENTIONS:
Behavioral: Family Spirit Nurture (FSN) — The FSN intervention will be conducted over a 6-month period. Participants in the intervention group will receive 6- 45 minute lessons in their home or a private place of their choosing. The lessons focus on elimination or reduction of Sugar Sweetened Beverages (SSBs) among infants while teaching mothers complementary feeding and responsive parenting practices
  Arms: Family Spirit Nurture (FSN)
Other: Control Program — The control group will receive three home-based lessons with home safety information.Lessons will be delivered monthly (at 3, 4 and 5 months postpartum) in the same format as the FSN lessons, by trained FHCs in the home of the participant or in a private place of their choosing.
  Arms: Control Program
Other: Water Delivery — Drinking water will be delivered to the household of each participant (both in the FSN intervention and control groups) from 6 to 9 months postpartum. The amount of water will be determined by the number of children and adults living in the household at the time of water delivery. The first delivery of water will occur at the time of the 6-month evaluation and the last delivery will occur at the time of the 9-month evaluation. Water will be delivered as often as weekly. Those families who do not need weekly water delivery (based on their preference and their usage of the first delivery of water) will receive water less frequently.

SUMMARY:
This study aims to assess the impact of a brief home-visiting module, called "Family Spirit Nurture" (FSN), on American Indian (AI) parent feeding practices associated with increased risk for early childhood obesity, with a primary focus on delaying introduction of infants' Sugar Sweetened Beverage (SSB) (including soda, energy drinks, juice with added sugar and other drinks with added sugar) intake while teaching mothers complementary feeding and responsive parenting practices. The investigators will also assess how water insecurity may moderate parents' feeding of SSBs to young children. Finally, the investigators will explore whether maternal knowledge of oral health practices and/or reduction of infants' SSB intake influences early indicators of infant's oral health (i.e., infants' oral microbiome and plaque formation). Our evaluation will employ a randomized controlled design, in which the control condition receives a beneficial home-safety educational model and assistance in safety proofing their homes for small children. Assessments in both groups will occur at baseline (between 6 and 10 weeks postpartum) and 4 months, 6 months, 9 months and 12 months postpartum.

Primary Aims:

Aim 1: To determine the effectiveness of the brief (6 lessons) FSN home-visiting parent feeding practice module on reducing SSB initiation and frequency among infants between 3 and 12 months of age. Hypothesis 1: Infants whose mothers receive FSN vs. controls will be less likely to introduce SSBs between 3 and 12 months of age.

Aim 2: To determine the effectiveness of FSN to promote optimal complementary feeding and responsive parenting practices. Hypothesis 2: Mothers who receive FSN vs. controls will be more likely to practice recommended complementary feeding and responsive parenting practices between 3 and 12 months of age.

Aim 3: To determine the impact of water insecurity on SSB consumption among infants between 3 and 6 months of age. Hypothesis 2: Parents who report water insecurity vs. those who do not will be more likely to give infants SSBs between 3 and 6 months of age.

Secondary Aims:

Secondary Aim 1: To explore if provision of water to families reduces SSB intake among mothers and infants ages 6 to 9 months of age.

Secondary Aim 2: To explore if infants in the FSN intervention have better oral health outcomes than control infants up to 12 months postpartum.

DETAILED DESCRIPTION:
The investigators will conduct a pilot randomized 1:1 controlled trial with 136 mother-infant dyads. Participants will be pre-screened for water insecurity and distributed equally across the two study arms using stratified block randomization. The intervention group (n=68) will receive the FSN home-visiting module, consisting of six 45-minute lessons delivered biweekly by trained local AI Family Health Coaches (FHCs), from 3 to 6 months postpartum. The lessons focus on elimination or reduction of Sugar Sweetened Beverages (SSBs) among infants while teaching mothers complementary feeding and responsive parenting practices. The control group (n=68) will receive three home-based lessons with home safety information (injury prevention is a priority identified by Navajo leadership that does not interfere with study questions). All families will receive delivery of drinking water from 6 to 9 months postpartum. Through this staggered design, the investigators will evaluate the impact of the FSN on infant feeding practices associated with increased risk for early childhood obesity, with a primary focus on delaying introduction of infant's SSB intake. The investigators will also be able to evaluate the impact of the availability of potable water on SSB intake, with or without family education. In addition, participants will have the opportunity to provide additional consent for a nested oral health study to evaluate the impact of the FSN curriculum and water provision on infant oral health indicators.

Methods:

Study implementation will include four phases:

Phase 1 (Referral, Recruitment, Consent, Baseline Assessment and Randomization): Potentially eligible mothers will be referred to our study staff, who will screen for eligibility, consent/assent mothers, conduct baseline assessment, and assign randomization status. Randomization will be assigned after the completion of the baseline assessment, including scoring of the participant's water insecurity status. Two randomization lists (one for water secure mothers and one for water insecure mothers) will be created prior to study initiation using STATA 14 statistical software37.

Part 2 (Home-Based Education Intervention): Local FHCs, trained and employed by Johns Hopkins, will deliver either the intervention (6-session FSN) or the control condition (3- Home-Safety Lessons) between 3 to 6 months postpartum.

Part 3 (Water Delivery): All participants will have drinking water delivered to their home from 6 to 9 months postpartum. FHCs will deliver water either weekly or less often, depending on needs of family. The amount of water delivered will be based on number of adults and children residing in home during this period of the study.

Part 4 (Assessment): Our assessment post-baseline consists of a mixed-methods assessment, including maternal self-reports and maternal FHC-administered interviews collected using REDCap at 4, 6, 7, 8, 9 and 12 months postpartum and maternal and infant medical chart reviews. If consent is given for the nested oral health study, the additional assessments will include a maternal self-report measure, collection and microbiologic testing of infant plaque and saliva, an infant oral examination, tooth eruption evaluations and infant medical and dental chart reviews.

ELIGIBILITY:
Inclusion Criteria:

1. American Indian ethnicity
2. Female
3. 13 years of age or older
4. Mother to a baby between the ages of 0 and 2.5 months
5. Living within 50 miles of the Northern Navajo Medical Center

Exclusion Criteria:

1. Inability to participate in full intervention or evaluation (e.g., planned move, residential treatment, etc.)
2. Unwilling to be randomized

Min Age: 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 136 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Reduction in SSB initiation and frequency among infants up to 12-months of age | 12-months of age
  To determine the effectiveness of the brief (6 lessons) FSN home-visiting parent feeding practice module on reducing SSB initiation and frequency among infants between 3 months and 12 months of age
Change in optimal complementary feeding and responsive parenting practices in mothers who receive FSN vs controls | 3-months and 12-months of age
  To determine the effectiveness of FSN to promote optimal complementary feeding and responsive parenting practices.
Change in SSB consumption among infants due to water insecurity | 6-months of age
  To determine the impact of water insecurity on SSB consumption among infants between 3 months and 6 months of age.

SECONDARY OUTCOMES:
Reduction in SSB intake among mothers and infants due to provision of water | 6-months to 9-months of age
  Explore if provision of water to families reduces SSB intake among mothers and infants
Change in oral health outcomes in infants in the FSN intervention vs control infants | Up to 12-months postpartum
  Explore if infants in the FSN intervention have better oral health outcomes than control infants

CONTACTS AND LOCATIONS:
Overall Officials: Allison Barlow, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Center for American Indian Health, Shiprock, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosenstock S, Ingalls A, Foy Cuddy R, Neault N, Littlepage S, Cohoe L, Nelson L, Shephard-Yazzie K, Yazzie S, Alikhani A, Reid R, Kenney A, Barlow A. Effect of a Home-Visiting Intervention to Reduce Early Childhood Obesity Among Native American Children: A Randomized Clinical Trial. JAMA Pediatr. 2021 Feb 1;175(2):133-142. doi: 10.1001/jamapediatrics.2020.3557. PMID 33165594